CLINICAL TRIAL: NCT06821477
Title: Impact of Knee Extension Brace on Quadriceps Electromyography Activity During Active Straight Leg Rise
Brief Title: Impact of Knee Extension Brace on Quadriceps EMG During ASLR
Status: Active, not recruiting | Type: Observational
Sponsor: Józef Piłsudski University of Physical Education (Other)
Responsible Party: Principal Investigator, Mateusz Kamiński, MSc PT, Józef Piłsudski University of Physical Education
Other Study IDs: EMG_brace
Record Dates: First submitted 2025-02-03; First posted 2025-02-12 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: EMG; Exercise Response

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 20 healthy young people: * age between 18-35 years
  * no contraindications to exercise
  * ability to perform the required commands without pain or discomfort
  * full range of motion of the knee joint.
  Interventions: Other: Superficial EMG

INTERVENTIONS:
Other: Superficial EMG — Superfiscial EMG during ASLR without knee brace follow by EMG during ASLR with knee brace under certain commands

SUMMARY:
The main objective of this study is to evaluate quadriceps thigh muscle activity during active straight leg raise (ASLR) with a knee brace.

An additional aim of the study is to evaluate quadriceps activity during straight leg raise with a knee brace in a variable command and manner of task performance. The study will be conducted on a group of healthy individuals aged 18 - 35 years. Height and weight were measured using a scale and centimetre tape. Then, according to the study protocol, specific measurements will be taken of the rectus femoris, medial vastus and lateral vastus muscles using surface EMG of a non-invasive nature.

Study participants will undergo the following measurements:

1. Measurement of the MVIC (maximum voluntary isometric contraction) of the quadriceps of the thigh, in a sitting position with the lower leg flexed to 90 degrees and in knee extended (0 degrees).
2. Measurement of muscle activity during elevation of the straightened lower limb in a supine position without an orthosis.
3. Measurement of muscle activity during straight leg raise in supine position with knee brace (default and different commends).

DETAILED DESCRIPTION:
The study will be conducted on a group of healthy individuals aged 18 - 35 years. After an interview confirming that the subject does not have exclusion criteria and inclusion criteria apply. Written consent to participate in the study and next anthropometric measurements will be taken using a scale and tape measure. The subjects will be informed in detail about the procedure and the form of the measurements, the way in which they are to be taken, and will be familiarized with the measuring instruments and their principles of operation. Then, in accordance with the study protocol, specific measurements will be taken of the rectus femoris, medial vastus and lateral vastus muscles using surface EMG of a non-invasive nature.

Study participants will undergo the following measurements:

1. Measurement of the MVIC (maximum voluntary isometric contraction) of the quadriceps femoris, in a sitting position with the lower leg flexed to 90 degrees, next MVIC of the quadriceps femoris in supine with knee fully extended (0 degrees).
2. Measurement of muscle activity during elevation of the straightened lower limb (ASLR) in supine without knee brace.
3. Measurement of muscle activity during ASLR in supine position with knee brace. Ad.a. Measurement of quadriceps maximum electric signal of the dominant lower limb using surface EMG in a seated position with the trunk stabilized with hands behind the pelvis and the lower leg flexed to 90 degrees, stabilized in the distal part (without taking the foot) against a stationary object (belt) to execute maximal volitional isometric quadriceps muscle contraction. Next MVIC in supine position, with knee fully extended, pushing back of the knee into hand of an examiner without lifting heel.

Ad.b. Measurement of quadriceps excitability using surface EMG in supine position without orthosis. The subject raises the tested limb (dominant) by touching the anterior surface of the tibia to a pole set at 30 cm at first sound of metronome set at 60 BMP, then hold the leg for the next beat, and next lowers the limb at the next metronome sound. This action is repeated three times in a row without any brake.

Ad.c. Measurement of quadriceps excitability of the dominant lower limb using surface EMG in supine position with knee extension brace on. Measurement performed in three variants:

1. The subject raises the test limb (dominant) by touching the anterior surface of the tibia to a pole set at 30 cm at first sound of metronome set at 60 BMP, then hold the leg for the next beat, and next lowers the limb at the next metronome sound. This action is repeated three times in a row without any brake.
2. The test subject is asked to apply maximum tension to the quadriceps then maintaining the tension he/she raises the limb touching the front surface of the tibia to the pole placed at the height of 30 cm at first sound of metronome set at 60 BMP, then hold the leg for the next beat, and next lowers the limb at the next metronome sound. This action is repeated three times.
3. Before the test, the test subject is verbally instructed to 'Try, despite the orthosis holding your knee straight, to bend the knee and raise the leg so that the quadriceps do not tense'. Then, lift the limb touching the front surface of the tibia to the pole placed at the height of 30 cm at first sound of metronome set at 60 BMP, then hold the leg for the next beat, and next lowers the limb at the next metronome sound. This activity is repeated three times.

Between MVICs and test trial it was 30s brake. MVICs were hold for 3 seconds. The time for the full test is approximately 15-20 minutes per participant. Statistical analysis will be performed using Statistica and/or JASP software. The study will be carried out with a minimum of 20 adults aged 18 - 35 years. The exact number of participants in the study, will be determined after performing an a-priori sample size estimation after collecting data from the first 10 people examined. Eligibility of subjects will include a subject and physical examination by a physiotherapist.

Inclusion criteria: age between 18-35 years, no contraindications to physical exercise, ability to perform the required commands without pain or discomfort, full range of motion of the knee joint.

Exclusion criteria: those with a history of knee and/or hip surgery, damage to ligamentous structures of the knee joint in the past treated conservatively or meniscus treated conservatively, muscle and tendon injury of the knee joint area in the past 3 months.

ELIGIBILITY:
Inclusion Criteria:

* age between 18-35 years
* no contraindications to exercise
* ability to perform the required commands without pain or discomfort
* full range of motion of the knee joint.

Exclusion Criteria:

* those with a history of knee and/or hip surgery
* damage to ligamentous structures of the knee joint in the past treated conservatively or meniscus treated conservatively.
* muscle and tendon injury of the knee joint area in the past 3 months.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: young healthy people 18-35 years old
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison between RF from p1 (ASLR without orthosis) to RF from p2 (ASLR with orthosis, without any command) | through study completion, an average of 1 year
  It was decided to choose RF and generalize it to whole quadriceps femoris, thus decide what is the impact of the extension brace on EMG quadriceps signal

SECONDARY OUTCOMES:
Muscle (RF, VLO, VMO) comparison between trials and inside every trial | through study completion, an average of 1 year
  Percentage of mean value from MVIC in 90 (standard EMG normalization), will be compared between trial (ex. p1 RF vs p2 RF vs p3 RF vs p4 RF) and inside each trial (ex. p1 RF vs p1 VLO vs p1 VMO).

OTHER OUTCOMES:
Comparison between analysis made with normalization to MVIC done in 90 degrees (standard) and done in 0 degrees (full extension). | through study completion, an average of 1 year
  Standard MVIC done on quadriceps muscle is done with knee bend to 90 degrees. We want to check what are the differences in analysis if the data will be normalized to MVIC done in 0 degrees.

CONTACTS AND LOCATIONS:
Locations (1):
- Jozef Pilsudski University of Physical Education, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD), including raw EMG data from electrodes and processed data normalized as %MVIC for statistical analysis, will be available upon reasonable request after primary results publication. Data will be anonymized to protect participant confidentiality and shared following ethical guidelines. Requests may be submitted to the corresponding author for up to 5 years post-publication.
Supporting Information: SAP, CSR
Access Criteria: Raw EMG data are available on reasonable request. We request investigators to contact us directly to discuss data sharing. On reasonable request statistical protocol and code for R or Python are available.